CLINICAL TRIAL: NCT03445533
Title: A Randomized Phase 3 Comparison of IMO-2125 With Ipilimumab Versus Ipilimumab Alone in Subjects With Anti-PD-1 Refractory Melanoma (ILLUMINATE-301)
Brief Title: A Study of Tilsotolimod in Combo With Ipilimumab vs Ipilimumab Alone in Subjects With Anti-PD-1 Refractory Melanoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2125-MEL-301
Record Dates: First submitted 2018-02-13; First posted 2018-02-26 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma; PD1; PD-1; refractory; metastatic; IMO-2125; illuminate 301; TLR9 agonist; advanced melanoma; CTLA4; CTLA-4; immunotherapy; skin cancer; ILLUMINATE-301
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Diabetes Mellitus, Insulin-Dependent, 12; Skin Neoplasms | interventions — Ipilimumab; tilsotolimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: ipilimumab (Experimental): ipilimumab 3 mg/kg intravenous
  Interventions: Drug: Ipilimumab
- Arm B: IMO-2125 plus ipilimumab (Experimental): IMO-2125 by intratumoral injection plus ipilimumab 3 mg/kg intravenous
  Interventions: Drug: Tilsotolimod with Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Arm A: 4 doses administered intravenously at a dose of 3 mg/kg over 90 minutes on Weeks 1, 4, 7, and 10.
  Other Names: Yervoy®
  Arms: Arm A: ipilimumab
Drug: Tilsotolimod with Ipilimumab — IMO-2125 intratumoral injection administered as 9 doses on Weeks 1, 2, 3, 5, 8, 11, 16, 20, and 24. WITH (Arm B): Ipilimumab administered as 4 doses on Weeks 2, 5, 8, and 11. in combination with tilsotolimod
  Other Names: IMO-2125 with Yervoy
  Arms: Arm B: IMO-2125 plus ipilimumab

SUMMARY:
A Phase 3 comparison of ipilimumab with and without IMO-2125 in advanced melanoma

DETAILED DESCRIPTION:
A Phase 3 global, multi-center, open-label comparison of ipilimumab with and without intratumoral IMO-2125 in subjects with advanced melanoma who had confirmed disease progression while on anti-PD-1

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing and able to sign the informed consent and comply with the study protocol.
2. Subjects must be ≥18 years of age.
3. Subjects must have histologically confirmed metastatic melanoma with measurable (by RECIST v1.1), stage III (lymph node or in transit lesions) or stage IVA, IVB, or IVC disease that is accessible for injection.
4. Patients must have confirmed progression during or after treatment with a PD-1 inhibitor (cannot be part of a bi-specific antibody) e.g. nivolumab or pembrolizumab. Confirmed progression is defined as:

   * Radiological progression (confirmed at least 4 weeks after the initial scan showing PD); or
   * (For progression based solely on worsening of non-target or new, non-measurable disease) confirmation by an additional scan at least 4 weeks after the initial scan unless it is accompanied by correlative symptoms.

   In addition, all the following must hold:
   1. No intervening anti-cancer therapy between the last course of PD-1 inhibitor treatment and the first dose of study treatment is allowed except for local measures (e.g., surgical excision or biopsy, focal radiation therapy).
   2. The interval between last PD-1 inhibitor and start of study treatment should be at least 21 days with no residual anti-PD-1-related immune toxicities in excess of Grade 1 severity.
   3. If BRAF mutation status is unknown, before randomization the subject must have BRAF testing performed using an approved assay method.
   4. Patients with BRAF-positive tumor(s) are eligible for the study if they received prior treatment with a BRAF inhibitor (alone of in combination with a MEK inhibitor) or declined targeted therapy.
5. Patients must have Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
6. Patients must meet the following laboratory criteria:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1500/mm3)
   2. Platelet count ≥ 75 x 10^9/L (75,000/mm3)
   3. Hemoglobin ≥ 8.0 g/dL (4.96 mmol/L)
   4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/minute
   5. Aspartate aminotransferase (AST) ≤ 2.5 x ULN; alanine aminotransferase (ALT) ≤ 2.5 x ULN; AST/ALT < 5 x ULN if liver involvement
   6. Serum bilirubin ≤ 1.5 x ULN, except in subjects with Gilbert's Syndrome who must have a total bilirubin < 3 mg/dL
7. Women of childbearing potential (WOCBP) and men must agree to use effective contraceptive methods from Screening throughout the study treatment period and until at least 90 days after the last dose of either ipilimumab or IMO-2125, whichever is later.
8. WOCBP must have a negative pregnancy test (serum or urine).

Exclusion Criteria:

1. Ocular melanoma.
2. Prior therapy with a toll-like receptor (TLR) agonist, excluding topical agents.
3. Prior ipilimumab treatment with the exception of adjuvant treatment completed ≥6 months prior to enrollment
4. Systemic treatment with interferon (IFN)-α within the previous 6 months.
5. Known hypersensitivity to any oligodeoxynucleotide.
6. Active autoimmune disease requiring disease-modifying therapy at the time of Screening.
7. Subjects requiring systemic steroid therapy receiving >10 mg/day of prednisone (or equivalent) for the 2 weeks preceding start of study.
8. Subjects with another primary malignancy that has not been in remission for at least 3 years, with the exception of non-melanoma skin cancer, curatively treated localized prostate cancer with non-detectable prostate-specific antigen, cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Papanicolaou (Pap) smear, and thyroid cancer (except anaplastic).
9. Active systemic infections requiring antibiotics
10. Active hepatitis A, B, or C infection.
11. Known diagnosis of human immunodeficiency virus (HIV) infection.
12. Women who are pregnant or breastfeeding.
13. Prior severe reaction to treatment with a human antibody that cannot be managed with standard supportive measures.
14. Presence of known central nervous system, meningeal, or epidural metastatic disease. However, subjects with known brain metastases are allowed if the brain metastases are stable for ≥4 weeks before the first dose of study treatment. Stable is defined as neurological symptoms not present or resolved to baseline, no radiologic evidence of progression, and steroid requirement of prednisone ≤10 mg/day or equivalent
15. Impaired cardiac function or clinically significant cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Idera Medical Director, Study Director — Idera Pharmaceuticals, Inc.
Locations (80):
- United States (16):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cancer Treatment Centers of America (CTCA) - Western Regional Medical Center, Scottsdale, Arizona
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Sutter Health Sacramento, Sacramento, California
  - University of California, San Diego (UCSD) - Moores Cancer Center, San Diego, California
  - Stanford Cancer Center, Stanford, California
  - Mount Sinai Medical Center of Florida, Inc., Miami Beach, Florida
  - University of Florida Health Cancer Center - Orlando Health, Orlando, Florida
  - The Valley Hospital, Ridgewood, New Jersey
  - University of Cincinnati Health, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center - Arthur G. James Cancer Hospital and Richard J. Solovev Research Institute (OSUCCC - James), Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Inova Health Care Services, Falls Church, Virginia
- Australia (6):
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Icon Cancer Center, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Queen Elizabeth Hospital, Woodville South, South Australia
  - University Hospital Geelong, Geelong, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Alberta Health Services Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Hopsital, Toronto, Ontario
- Czechia (3):
  - Fakultni nemocnice Olomouc - Oncology clinic, Olomouc
  - Dermatovenerologika Klinika, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (12):
  - CHU - Clermont Ferrand, Clermont-Ferrand, Cedex
  - CHRU Besançon - Jean Minjoz, Rouen, Cedex
  - CHU Amiens Picardie - Hopital Sud, Amiens
  - CHU Dijon - Hôpital Mitterrand, Dijon
  - CHU de Grenoble, La Tronche
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - Centre Leon Berard, Lyon
  - CHU de Marseille - Hopital de la Timone, Marseille
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Hopitaux de Rouen, Rouen
  - Institut Gustave Roussy, Villejuif
- Germany (9):
  - Klinikum Augsburg, Augsburg
  - Charite Universitaetsmedizin Berlin, Berlin
  - Elbe Kliniken, Buxtehude
  - Medizinische Hochschule Hannover - Klinik for Dermatologie, Allergologie und Venerologie, Hannover
  - Universitaetsklinikum Heidelberg Universitaets-Hautklinik, Heidelberg
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Universitatsklinikum Regensburg, Regensburg
  - Universität Tübingen, Tübingen
  - Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Universität Würzburg, Würzburg
- Italy (13):
  - Azienda Ospedale Policlinico di Bari, Bari
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico Bari, Bari
  - ASST degli Spedali Civili di Brescia, Brescia
  - IRCCS Azienda Ospedaliera Universitaria San Martino IST, Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Istituto Nazionale di Tumori IRCCS "Fondazione Sen. G. Pascale", Napoli
  - Istituto Oncologico Veneto-I.R.C.C.S., Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Azienda Ospedaliero Universitaria Senese, Siena
  - Universita di Torino, Torino
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (10):
  - Hospital Universitario A Coruna, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Quiron Dexeus Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Onkologikoa, Donostia / San Sebastian
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Consorci Hospital General Universitari de Valencia, Valencia
- Sweden (3):
  - Skånes Universitetssjukhus i Lund, Lund
  - Karolinska Universitetssjukhuset, Solna
  - Centrallasarettet i Växjö, Vaxjo
- United Kingdom (3):
  - Bristol Haematology and Oncology Centre, Bristol
  - Guy's Hospital, London
  - Royal Marsden Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diab A, Ascierto PA, Maio M, Abdel-Wahab R, Negrier S, Mortier L, Arenberger P, Dalle S, Krajsova I, de la Cruz L, Leccia MT, Guida M, Lebbe C, Grob JJ, Butler MO, In GK, Loquai C, Walker JWT, Atkinson V, Kapiteijn E, Haferkamp S, Chunduru S, Rahimian S, Guidoboni M, Robert C. Randomized, Open-Label, Phase III Study of Tilsotolimod in Combination With Ipilimumab Versus Ipilimumab Alone in Patients With Advanced Refractory Melanoma (ILLUMINATE-301). J Clin Oncol. 2025 May 20;43(15):1800-1809. doi: 10.1200/JCO.24.00727. Epub 2025 Mar 6. PMID 40048691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The global Phase 3 study was conducted at academic cancer centers across 11 countries. Participating countries included United States, Australia, Canada, Czech Republic, France, Germany, Italy, Netherlands, Spain, Sweden, and United Kingdom.
Pre-assignment Details: The study was an open-label comparison of ipilimumab with and without intratumoral IMO-2125 (tilsotolimod) in participants with advanced melanoma who had disease progression while on or after PD-1 directed therapy. Study participants were randomized 1:1 to ipilimumab alone (Arm A) or ipilimumab with tilsotolimod given intratumorally (Arm B). Randomization was stratified on the duration of prior anti-PD-1 therapy, metastasis stage, and BRAF mutation status.
Groups:
- Arm B: IMO-2125 (Tilsotolimod) Plus Ipilimumab: IMO-2125 by intratumoral injection plus ipilimumab 3 mg/kg intravenous
  Tilsotolimod with ipilimumab: IMO-2125 intratumoral injection administered as 9 doses on Weeks 1, 2, 3, 5, 8, 11, 16, 20, and 24. WITH (Arm B): Ipilimumab administered as 4 doses on Weeks 2, 5, 8, and 11. in combination with tilsotolimod.
Period: Overall Study
Arm/Group | Arm A: Ipilimumab | Arm B: IMO-2125 (Tilsotolimod) Plus Ipilimumab
Started | 243 | 238
Completed | 115 | 45
Not Completed | 128 | 193
Not completed — Progressive Disease | 48 | 81
Not completed — Adverse Event | 60 | 64
Not completed — Death | 9 | 19
Not completed — Miscellaneous | 0 | 16
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Physician Decision | 1 | 3
Not completed — Sponsor Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Never Received any Study Treatment | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Ipilimumab | Arm B: IMO-2125 Plus Ipilimumab | Total
Number analyzed (Participants) | 243 | 238 | 481
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (13.73) | 64.3 (13.28) | 64.3 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 105 | 221
  Male | 127 | 133 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 211 | 187 | 398
  Unknown or Not Reported | 27 | 45 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 207 | 187 | 394
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 27 | 44 | 71
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 9 | 11 | 20
  Netherlands | 9 | 2 | 11
  Sweden | 2 | 3 | 5
  United States | 23 | 23 | 46
  Czechia | 11 | 19 | 30
  Italy | 53 | 40 | 93
  United Kingdom | 2 | 3 | 5
  Australia | 10 | 4 | 14
  France | 71 | 97 | 168
  Germany | 24 | 14 | 38
  Spain | 29 | 22 | 51
Baseline Melanoma Characteristics [Count of Participants; unit: Participants]
  Primary Histology - Cutaneous | 210 | 203 | 413
  Primary Histology - Mucosal | 14 | 12 | 26
  Primary Histology - Other | 18 | 23 | 41
  Primary Histology - Missing | 1 | 0 | 1
Baseline Melanoma Staging [Count of Participants; unit: Participants] — Measure Description: Physician assessed and determined based on American Joint Committee on Cancer (AJCC) Staging System for Melanoma, Seventh Edition, which determines the stage (I-V) based on the TNM classification. T refers to tumor size, N refers to nearby lymph nodes and M represents metastasized (spread) to other parts of the body. This staging number is obtained as a sum of the TNM classification. The lower the number, the lower the cancer stage and the better the prognosis for the patient. The higher the stage, the worse the prognosis for the patient.
  Participants
    IIIA | 0 | 1 | 1
    IIIB | 0 | 2 | 2
    IIIC | 20 | 35 | 55
    IVM1A | 36 | 24 | 60
    IVM1B | 46 | 24 | 70
    IVM1C | 137 | 147 | 284
    Other | 4 | 5 | 9
Baseline Elevated LDH (lactate dehydrogenase) [Count of Participants; unit: Participants]
  Yes | 124 | 126 | 250
  No | 112 | 106 | 218
  Unknown | 7 | 6 | 13
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status Scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). Scale grades are from 0 (fully active) best to 5 (dead) worst and are determined by physician assessment of the patient.
  Grade:
  0 - Fully active
  1. - Restricted in physically strenuous activity
  2. - Ambulatory, but unable to work
  3. - Limited selfcare, confined to bed/chair > 50% of waking hours
  4. - Completely disabled, confined to bed/chair, no selfcare
  5. - Dead
  Participants
    0 | 146 | 150 | 296
    1 | 96 | 87 | 183
    2 | 1 | 1 | 2
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
    5 | 0 | 0 | 0
Prior Systemic Anti-cancer Treatment [Number; unit: Prior Treatments] — Indicates multiple, known treatments. Participants may be counted in more than one category based on the combination of prior treatments.
  Prior Treatments
    PD-1 Inhibitor | 242 | 237 | 479
    BRAK Inhibitor | 36 | 35 | 71
    MEK Inhibitor | 36 | 33 | 69
    Other | 27 | 38 | 65
    Other Immunotherapy | 14 | 18 | 32
    Cytokine | 14 | 10 | 24
    Chemotherapy | 8 | 11 | 19
    CTLA-4 Inhibitor | 5 | 6 | 11
    Oncolytic Virus | 6 | 5 | 11
    Other Targeted Therapy | 6 | 5 | 11
Prior Systemic Anti-cancer Treatment Setting [Number; unit: Prior Treatment Settings]
  Unresectable/Metastatic Disease | 214 | 200 | 414
  Adjuvant | 58 | 76 | 134
  Neoadjuvant | 6 | 2 | 8
  Other | 1 | 4 | 5
Best Response from Last Prior Systemic Anti-cancer Treatment [Count of Participants; unit: Participants]
  Complete Response | 6 | 3 | 9
  Partial Response | 26 | 23 | 49
  Stable Disease | 49 | 49 | 98
  Progressive Disease | 135 | 125 | 260
  Unknown | 27 | 38 | 65
Duration of Prior Anti-PD-1 Therapy [Count of Participants; unit: Participants]
  Greater than or Equal to 12 Weeks | 207 | 204 | 411
  Less than 12 Weeks | 36 | 34 | 70
BRAF Mutation Status and Prior Targeted Therapy [Count of Participants; unit: Participants]
  BRAF Wild Type | 188 | 186 | 374
  BRAF Mutation Positive with Prior Targeted Therapy | 35 | 34 | 69
  BRAF Mutation Positive with no Prior Targeted Therapy | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Summary of Independent Reviewer-Assessed Objective Response Rate (ORR) by RECIST v1.1
Description: The ORR for evaluable participants was calculated using the participant's best overall response (BOR).
  Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for target lesions as assessed by MRI, CT or X-ray: Complete Response (CR) - disappearance of all target lesions; Partial Response (PR) - >=30% decrease from baseline of the sum of diameters of all target lesions; Stable Disease (SD) - does not qualify for CR, PR or Progression; Progressive Disease (PD) - 20% increase in the sum of diameters of target lesions.
  The calculation is derived from measuring the diameter (mm) of the target lesion at baseline and comparing target lesion diameter (mm) at intervals during treatment and/or post-treatment. Based on the percent of tumor decrease or increase, the appropriate category is assigned.
Time Frame: Response is measured from the date of randomization, until disease progression, death, or start of new anti-cancer therapy (up to 36 months).
Population: All percentages were based on the number of participants in the Intent-to-Treat (ITT) analysis set within each group. Participants with no disease assessment in the study were included in the Not Evaluable category under Best Overall Response.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ipilimumab | Arm B: IMO-2125 Plus Ipilimumab
Number analyzed (Participants) | 243 | 238
Participants
  Complete Response | 1 | 1
  Partial Response | 20 | 20
  Stable Disease | 45 | 61
  Progressive Disease | 110 | 89
  Not Evaluable | 67 | 67
Statistical Analysis 1: Comparison: Arm A: Ipilimumab vs Arm B: IMO-2125 Plus Ipilimumab; The ORR was defined as a percentage of subjects meeting criteria of CR and PR to calculate the p-value; Test type: Superiority; p = 0.9394, Cochran-Mantel-Haenszel — p-value was calculated for percentage difference (B-A) using a Cochran-Mantel-Haenszel (CMH) test stratified by metastasis stage and BRAF mutation; ORR and OS comprise a primary endpoint family; both have a priori hypotheses and were tested for statistical significance

2. Primary Outcome: Summary of Overall Survival
Description: Efficacy measured by overall survival (OS) was defined as the number of participants alive compared to the number of participants that died by treatment group.
Time Frame: OS is measured from the date of randomization to the date of death from any cause (up to 36 months).
Population: All percentages were based on the number of participants in the Intent-to-Treat (ITT) analysis set within each group.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ipilimumab | Arm B: IMO-2125 Plus Ipilimumab
Number analyzed (Participants) | 243 | 238
Participants
  Died | 166 | 165
  Alive (Censored) | 77 | 73
Statistical Analysis 1: Comparison: Arm A: Ipilimumab vs Arm B: IMO-2125 Plus Ipilimumab; Test type: Superiority; p = 0.6775, Log Rank — The p-value was calculated using the log rank test stratified by metastasis stage and BRAF mutation; ORR and OS comprise a primary endpoint family; both have a priori hypotheses. ORR will be tested first followed by OS; Cox Proportional Hazard = 0.955, 95% CI 2-sided [0.770 to 1.186] — Hazard ratio and 95% CI (B/A) are estimated using a Cox proportional hazards model stratified by metastasis stage and BRAF mutation

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signing of informed consent, through the duration of active study treatment (10 weeks active study for participants assigned to Arm A OR 24 weeks active study for participants assigned to Arm B) and then for 90 days after the last dose of study treatment. All-Cause Mortality was assessed for up to 36 months.
Description: Definitions aligned with FDA and ICH requirements.
  The grading of adverse events utilized the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03, which were defined as:
  Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening, and Grade 5 = Death
Arm/Group | Arm A: Ipilimumab | Arm B: IMO-2125 (Tilsotolimod) Plus Ipilimumab
All-Cause Mortality (participants affected / at risk) | 166/243 | 165/238
Serious Adverse Events (participants affected / at risk) | 108/243 | 119/238
Other Adverse Events (participants affected / at risk) | 218/243 | 226/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Ipilimumab (N=243) | Arm B: IMO-2125 (Tilsotolimod) Plus Ipilimumab (N=238)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Lymph Node Pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 2 (5)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular Disorder (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Immune-mediated Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 6 (7) | 3 (3)
Adrenal Insufficiency (Endocrine disorders) | 3 (3) | 2 (2)
Adrenocortical Insufficiency Acute (Endocrine disorders) | 0 (0) | 1 (1)
Adrenocorticotropic Hormone Deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Lymphocytic Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 13 (17) | 10 (10)
Immune-mediated Enterocolitis (Gastrointestinal disorders) | 11 (13) | 11 (14)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Autoimmune Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Toxicity (Gastrointestinal disorders) | 1 (1) | 1 (1)
Immune-mediated Pancreatitis (Gastrointestinal disorders) | 1 (3) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (2) | 0 (0)
Chronic Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gingival Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedematous Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 8 (10) | 12 (17)
General Physical Health Deterioration (General disorders) | 5 (5) | 6 (8)
Asthenia (General disorders) | 3 (3) | 2 (2)
Influenza Like Illness (General disorders) | 1 (1) | 2 (2)
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Ill-Defined Disorder (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 0 (0)
Immune-mediated Hepatitis (Hepatobiliary disorders) | 5 (5) | 6 (8)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 3 (3)
Cholestasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Autoimmune Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular Injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 4 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 4 (5)
Cytokine Release Syndrome (Immune system disorders) | 0 (0) | 3 (3)
Anaphylactoid Reaction (Immune system disorders) | 0 (0) | 1 (1)
Haemophagocytic Lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 5 (5) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 4 (5)
Cellulitis (Infections and infestations) | 3 (4) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Dermo-hypodermitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Abdominal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis Viral (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis Streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Groin Abscess (Infections and infestations) | 1 (1) | 0 (0)
Injection Site Abscess (Infections and infestations) | 0 (0) | 1 (1)
Injection Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Aseptic (Infections and infestations) | 1 (2) | 0 (0)
Oesophageal Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Parvovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 (0) | 1 (1)
Post Procedural Infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injection Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 0 (0)
Troponin Increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperglycaemic Hyperosmolar nonketotic Syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Intracranial Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Infected Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin Neoplasm Bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour Necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Central Nervous System Necrosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-barre Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Limbic Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transverse Sinus Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Immune-mediated Nephritis (Renal and urinary disorders) | 1 (1) | 1 (1)
Autoimmune Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis Hemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Immune-mediated Renal Disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (6)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Jugular Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Ipilimumab (N=243) | Arm B: IMO-2125 (Tilsotolimod) Plus Ipilimumab (N=238)
Anaemia (Blood and lymphatic system disorders) | 31 (57) | 37 (61)
Diarrhoea (Gastrointestinal disorders) | 61 (85) | 70 (108)
Nausea (Gastrointestinal disorders) | 48 (56) | 54 (67)
Vomiting (Gastrointestinal disorders) | 30 (35) | 35 (40)
Constipation (Gastrointestinal disorders) | 23 (24) | 21 (23)
Abdominal Pain (Gastrointestinal disorders) | 13 (14) | 21 (24)
Dry Mouth (Gastrointestinal disorders) | 13 (13) | 13 (14)
Abdominal Pain Upper (Gastrointestinal disorders) | 15 (17) | 8 (8)
Asthenia (General disorders) | 52 (60) | 79 (110)
Pyrexia (General disorders) | 28 (42) | 102 (211)
Fatigue (General disorders) | 35 (44) | 48 (75)
Chills (General disorders) | 7 (7) | 75 (120)
Influenza Like Illness (General disorders) | 5 (7) | 30 (61)
Injection Site Pain (General disorders) | 0 (0) | 22 (30)
Hepatocellular Injury (Hepatobiliary disorders) | 8 (11) | 14 (15)
Cholestasis (Hepatobiliary disorders) | 5 (6) | 13 (14)
Aspartate Aminotransferase Increased (Investigations) | 18 (25) | 32 (54)
Alanine Aminotransferase Increased (Investigations) | 18 (27) | 31 (51)
Weight Decreased (Investigations) | 12 (15) | 25 (33)
Blood Alkaline Phosphate Increased (Investigations) | 8 (9) | 16 (19)
Gamma-glutamyltransferase Increased (Investigations) | 3 (5) | 16 (23)
Decreased Appetite (Metabolism and nutrition disorders) | 42 (46) | 45 (49)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (16) | 18 (26)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (8) | 14 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (20) | 18 (24)
Back Pain (Musculoskeletal and connective tissue disorders) | 17 (18) | 12 (12)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 12 (13) | 11 (13)
Headache (Nervous system disorders) | 15 (20) | 43 (60)
Insomnia (Psychiatric disorders) | 14 (14) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 19 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 17 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 60 (70) | 57 (72)
Rash (Skin and subcutaneous tissue disorders) | 22 (32) | 22 (30)
Vitiligo (Skin and subcutaneous tissue disorders) | 3 (4) | 15 (17)
Erythema (Skin and subcutaneous tissue disorders) | 5 (6) | 12 (14)
Hypotension (Vascular disorders) | 0 (0) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT03445533/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT03445533/SAP_001.pdf